CLINICAL TRIAL: NCT04910113
Title: Bronchiectasis as Atypical Presentation in COVID-19: A Single Center Study
Brief Title: Bronchiactasis as Atypical Presentation in COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Ahmed Abd El-Gawad Mohamed Okash, Principal investigator, Assiut University
Other Study IDs: COVID in Bronchiactasis
Record Dates: First submitted 2021-05-17; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Covid19 in Bronchiactasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the prevelance and pattern of bronchiectasis as atypical COVID-19 presentation

DETAILED DESCRIPTION:
bronchiectasis is achronic inflammatory lung disease. It is defined by the presence of permanent and abnormal dilatation of the bronchi. which leads to chronic sputum production and impaired bacterial clearance. The affected parts of the lungs develop a vicious cycle of failed pathogen clearance leading to frequent infections, chronic inflammation and ongoing structural damage. The main symptoms are daily cough, daily sputum production and frequent respiratory infections. There is low frequency of non cystic fibrosis bronchiectasis The prevalence rate of NCFB in the general population was calculated to be 39.9 cases per 100,000.

There is an increasing prevalence of bronchiectasis in the elderly, affecting approximately 10 patients per 1,000 population.

A retrospective cohort study of health claims between 1999-2001 in the US suggested the prevalence of bronchiectasis to be 4.2 per 100,000 population aged 1834 years and 271.8 per 100,000 population aged >75 years . This usually occurs in the context of chronic airway infection causing inflammation. The main clinical manifestation is a productive cough. Bronchiectasis is currently nearly always diagnosed using high-resolution computed tomography (HRCT) scanning. The main diagnostic features are: 1) internal diameter of a bronchus is wider than its adjacent pulmonary artery; 2) failure of the bronchi to taper; and 3) visualization of bronchi in the outer 12 cm of the lung fields.

Coronaviruses (CoVs) are a group of highly diverse, enveloped, positive-sense, and single-stranded RNA viruses.

In late December 2019, an outbreak of an unknown disease called pneumonia of unknown cause occurred in Wuhan, Hubei province, China.1 The outbreak has spread substantial to infect 9720 people in China with 213 deaths and to infect 106 people in 19 other countries up to 31 January 2020 . A few days later, the causative agent of this mysterious pneumonia was identified as a novel coronavirus (nCoV) by several independent laboratories.2-4 The causative virus has been temporarily named as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the relevant infected disease has been named as coronavirus disease 2019 (COVID-19) by the World Health Organization, respectively. According to the daily report of the World Health Organization, the epidemic of SARS-CoV-2 so far registered 78630 cases and 2747 deaths in China, spread to 46 other countries that reported a total of 3664 cases by 27 February 2020 . COVID-19 epidemic has become a global health threat. Coronaviruses (CoVs) are a group of highly diverse, enveloped, positive-sense, and single-stranded RNA viruses.5 They cause several diseases involving respiratory, enteric, hepatic, and neurological systems with vary severity among humans and animals.6,7 The envelope spike (S) protein is important for CoV.19 The S protein mediates receptor binding and membrane fusion and is crucial for determining host tropism and transmission capacity.8,9,10 The final etiologic diagnosis of COVID-19 is nessary can be farther further confirmed with a positive real-time RT-PCR assay for COVID-19 using respiratory or blood samples or by means of viral gene sequencing of respiratory or blood samples that are highly homologous with COVID-19.

The typical chest CT findings include multifocal bilateral ground-glass opacities (GGOs) with patchy consolidations, prominent peripherally subpleural distribution, and posterior part or lower lobe predilection.

The long-term sequelae of COVID-19 remain to be investigated, although several publications have reported a fibrotic phase with reticulation characteristics, interlobar septal thickening, and traction bronchiectasis.

The onset and development of bronchiectasis during the follow-up of COVID-19 patients with pneumonia are under-reported.

ELIGIBILITY:
Inclusion Criteria:

* Significant sputum production (≥ 10 ml per day)
* Adult patients aged 18 years or older of both sex and diagnosed as COVID-19 positive by PCR either during same visit or in previous visits during the 2020-2021 who have CT scan examination of the chest during acute diseases or at follow up

Exclusion Criteria:

* Children under 18 years old, patients with known chronic chest diseases, and patients who are not examined by CT scan of the chest

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Includes all patients admitted to Assuit police hospital diagnosed as COVID-19 positive by PCR and meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of bronchiectasis among COVID-19 patients | 1year
  To evaluate the prevelance and pattern of bronchiectasis as atypical COVID-19 presentation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shaddad, Lecture, Principal Investigator — Assuit University - Assuit - Egypt
Locations (1):
- Maha Ahmed Okasha, Asyut, Egypt